CLINICAL TRIAL: NCT05353205
Title: A Double-blind , Randomized, Multicenter, Phase 4 Study to Evaluate Efficacy and Safety of Oral Flumatinib 400mg Versus 600mg in Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase.
Brief Title: A Study of the Efficacy and Safety of Flumatinib in Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10096-402
Record Dates: First submitted 2022-04-22; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: CML, Chronic Phase
Keywords: CML, Chronic Phase; Flumatinib; BCR-ABL TKI; Dose-optimization; Double-blind; Phase 4
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flumatinib (400mg) (Experimental): Flumatinib 400mg QD
  Interventions: Drug: Flumatinib mesylate tablets (400mg)
- Flumatinib (600mg) (Experimental): Flumatinib 600mg QD
  Interventions: Drug: Flumatinib mesylate tablets (600mg)

INTERVENTIONS:
Drug: Flumatinib mesylate tablets (400mg) — Flumatinib 400mg +Placebo for flumatinib are administered orally daily. Patients are randomized to flumatinib 400mg QD.
  Arms: Flumatinib (400mg)
Drug: Flumatinib mesylate tablets (600mg) — Flumatinib 600mg is administered orally daily. Patients are randomized to flumatinib 600mg QD.
  Arms: Flumatinib (600mg)

SUMMARY:
It's a double-blind , randomized ,multi-center study. The purpose of this study is to explore the efficacy and safety of flumatinib 400mg once daily (QD) versus 600mg QD as the first line therapy in patients with chronic myleiod leukemia(CML) in chronic phase(CP).

DETAILED DESCRIPTION:
This is a dose-optimization study of flumatinib in adult patient with newly diagnosed CML-CP. The objective of this study is to compare the efficacy and safety of flumatinib 400mg QD with that of 600mg QD. Eligible patients are randomized in a 1:1 ratio to receive either fluamtinib 400mg QD or flumatinib 600mg QD. Randomization is stratified based on Sokal risk score (<0.8,0.8~1.2,>1.2). Patients will discontinue study therapy due to treatment failure, disease progression or intolerance to study medication or due to investigator's or participant's decision. The primary efficacy endpoint is the rate of early molecular response , as measured by RQ-PCR at 3 months. Hematologic response, molecular response and cytogenetic response will be assessed at baseline and a certain frequency after treatment, until study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Men or women aged more than or equal to (≥) 18 years, and less than (<) 75 years.
3. ECOG performance status of 0-2.
4. Patients with philadelphia chromosome positive chronic myeloid leukemia in chronic phase (Ph+ CML-CP) within 6 months of diagnosis.
5. Adequate organ function.
6. Men or women should be using adequate contraceptive measures throughout the study; Females should not be breastfeeding at the time of screening, during the study and until 6 months after completion of the study.
7. Females must have evidence of non-childbearing potential.

Exclusion Criteria:

1. Known atypical CML or presence of additional chromosomal abnormalities.
2. Known presence of the T315I mutation.
3. Treatment with tyrosine kinase inhibitor(s) prior to randomization.
4. Any treatment with anti-CML activity for longer than 2 weeks(exception of hydroxyurea or anagrelide) or hematopoietic stem cell transplantation prior to randomization .
5. Prior treatment with splenectomy.
6. Impaired cardiac function including any one of the following:

   1. Resting corrected QT interval (QTc) > 470 ms obtained from electrocardiogram (ECG), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG.
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events,
   4. Left ventricular ejection fraction (LVEF) ≤ 50%.
   5. During screening period, ECG examination showed average heart rate <50 beats per minute.
   6. Myocardial infarction occurred within 12 months of randomization;
   7. Congestive heart failure occurred within 6 months of randomization;
   8. Uncontrollable angina.
7. Stroke or transient ischemic attack within 6 months of randomization.
8. Any severe or uncontrolled systemic diseases (i.e. uncontrolled hypertension or diabetes).
9. Clinically severe gastrointestinal dysfunction that may affect drug intake, transport or absorption.
10. The presence of active infectious diseases has been known prior to randomization
11. History of significant congenital or acquired bleeding disorders unrelated to CML
12. Inadequate other organ function.
13. History of other malignancies.
14. History of hypersensitivity to any active or inactive ingredient of flumatinib.
15. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued.
16. Major surgery within 4 weeks of randomization.
17. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 within 4 weeks of randomization.
18. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.
19. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Early molecular response(EMR) rate at 3 months | 3 months
  Molecular response is assessed using BCR-ABL transcript levels and measured by realtime quantitative polymerase chain reaction(RQ-PCR). Early molecular response is defined as a ratio BCR-ABL/ABL ≤10% on the international scale (IS).

SECONDARY OUTCOMES:
Major molecular response(MMR) rate at month 3,6,9 and 12 | 3, 6, 9 and 12 months
  Major molecular response is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale as measured by RQ-PCR.
MR4.0 rate at month 3,6,9 and 12 | 3, 6, 9 and 12 months
  MR4.0 is defined as BCR-ABL/ABL ≤0.01% on the international scale.
MR4.5 rate at month 3,6,9 and 12 | 3, 6, 9 and 12 months
  MR4.5 is defined as BCR-ABL/ABL ≤0.0032% on the international scale.
Complete cytogenetic response（CCyR）rate at month 3,6,9 and 12 | 3, 6, 9 and 12 months
  Cytogenetic response (CyR) is based on the prevalence of Ph+ cells in metaphase from bone marrow (BM) sample . CCyR is defined as 0% Ph+ metaphases in the bone marrow.
Complete hematologic response(CHR) rate at month 1,2,3,4,5,6,9 and 12 | 1,2,3,4,5,6,9 and 12 months
  Hematologic response will be assessed by complete blood count (CBC) and physical examination at each visit. CHR is defined as all of the following present:
  1. white blood cell(WBC) count <10×109/L
  2. Platelet count <450 ×109/L
  3. Peripheral blood basophils <5%
  4. No blasts and no promyelocytes in peripheral blood
  5. < 5% myelocytes plus metamyelocytes in peripheral blood
  6. No evidence of extramedullary disease, including no splenomegaly or hepatomegaly
Time to first MMR | up to 36 months
  Evaluate the time from the date of randomization to the date of first documented MMR during treatment.
Time to first CCyR | up to 36 months
  Evaluate the time from the date of randomization to the date of first documented CCyR during treatment.
Duration of MMR | up to 36 months
  Duration of MMR is defined as the time from the date of first documented MMR to the earliest date of loss of MMR.
Duration of CCyR | up to 36 months
  Duration of CCyR is defined as the time from the date of first documented CCyR to the earliest date of loss of CCyR.
Event-free survival (EFS) | up to 36 months
  EFS is defined as the time from the date of randomization to the earliest occurrence of the following events: death due to any cause ; loss of CHR ,loss of PCyR ;loss of CCyR ; discontinuation of study treatment due to AE or treatment failure ; progression to AP/BC
Progression-free survival (PFS) | up to 36 months
  PFS is defined as the time from the date of randomization to the earliest occurrence of progression to AP/BC or death from any cause.
Overall survival (OS) | Frame:12 and 36 months
  OS is defined as the time from the date of randomization to the date of death from any cause.
The incidence and severity of adverse events ((AE) | up to 36 months
  Assessed by number and severity of adverse events as recorded on the case report form NCI CTCAE v5.0.
Pharmacokinetics (PK) of HS-10096：Tmax | Up to approximately 36 months
  Serum concentrations of HS-10096 will be collected and analyzed to evaluate the PK of HS-10096.Tmax is the time to reach maximum (peak) plasma drug concentration after dose administration (hr).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — Institute of Hematology and Oncology, Harbin The First Hospital
Locations (1):
- Institute of Hematology and Oncology, Harbin The First Hospital, Harbin, Hei Longjiang, China